CLINICAL TRIAL: NCT04876053
Title: Home Food Delivery for Diabetes Management in Patients of Rural Clinics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 261074
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Diet, Healthy
Keywords: Food Insecurity
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention)
- Healthy Food Delivery Intervention (Experimental): 9000 calorie / week food box
  Interventions: Behavioral: Healthy Food Delivery Intervention

INTERVENTIONS:
Behavioral: Healthy Food Delivery Intervention — Each weekly food box will include ~9,000 calories of food, equivalent to the amount the average household receives prorated per week from an average Arkansas food pantry. The boxes will be designed by a registered dietitian. The boxes will follow ADA's Create Your Plate method consistent with the meal pattern promoted in the American College of Physicians (ACP) DSMES. The foods will also reflect Feeding America's Detailed Foods to Encourage framework, developed by nutrition experts and food bank staff to represent USDA dietary guidelines with healthy food that can be made available by food banks.
  Arms: Healthy Food Delivery Intervention

SUMMARY:
Our long-term goal is to transform rural residents' management of T2DM. This study's objective is to determine the effectiveness of an intervention that is scalable and sustainable and promotes patient adherence by mitigating rural food insecure participants' difficulties associated with completing existing interventions. Our specific aims are:

1. Compare the effectiveness of the Healthy Food Delivery Intervention (HFDI) plus standard care and standard care alone to improve diabetes-related outcomes among rural food insecure patients with T2DM. Hypothesis: Compared with standard care alone, patients receiving the HFDI plus standard care will demonstrate improved: H1 glycemic control as measured by HbA1c; H2 cardio-metabolic risk factors: blood pressure, fasting glucose, fasting lipids, and BMI; H3 self-management: self-efficacy, adherence to self-management behaviors, and medication adherence; H4 patient-centered outcomes: diabetes-related distress, diabetes-related quality of life, and diabetes-related complications.
2. Compare the effectiveness of the HFDI plus standard care and standard care alone to improve diet quality among rural food insecure patients with T2DM. Hypothesis: Compared with standard care alone, patients receiving the HFDI plus standard care will demonstrate improved: H1 Healthy Eating Index 2015 (HEI-2015) scores; H2 fruit and vegetable consumption.
3. Compare cost-effectiveness to understand HFDI plus standard care costs in relationship to outcomes in relation to standard care alone. Hypothesis: The HFDI will be cost-effective based on traditional cost per additional quality-adjusted life year gained.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* report food insecurity
* report T2D (confirmed by having an HbA1c equal to or greater than 6.5 at initial data collection immediately following consent)
* Speak English or Spanish
* Currently lives at a rural address

Exclusion Criteria:

* conditions making it unlikely the participant will be able to follow the protocol, such as terminal illness, severe mental illness, severely impaired vision or hearing, eating disorder, or plans to move out of the geographic region
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline to immediate post-intervention (approx. 18 weeks)
  Finger stick blood collection will be used to test HbA1c using a Siemens DCA Vantage.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Long, PhD, Principal Investigator — University of Arkansas
Locations (4):
- United States (4):
  - UAMS - North Central, Batesville, Arkansas
  - UAMS - East, Helena, Arkansas
  - UAMS - Northeast, Jonesboro, Arkansas
  - UAMS - South, Magnolia, Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Short E, Selig JP, Felix HC, Painter J, McElfish PA, Rowland B, Ammerman AS, Bounds K, Henske J, Hudson JS, Li J, Young SG, Long CR. Healthy food delivery for type 2 diabetes management in rural clinics' patients: A comparative effectiveness randomized controlled trial protocol. Contemp Clin Trials. 2024 May;140:107491. doi: 10.1016/j.cct.2024.107491. Epub 2024 Mar 6. PMID 38458560

DOCUMENTS (1):
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04876053/ICF_000.pdf